CLINICAL TRIAL: NCT00551382
Title: Phase 3 Study of Montelukast as Prophylaxis for Upper Respiratory Tract Infections in Children
Brief Title: Montelukast as Prophylaxis for Upper Respiratory Tract Infections in Children: a Randomised, Double-blind, Placebo-controlled Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Berkovitch M, Assaf Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 142/06; 20060504(142/06)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Upper Respiratory Tract Infection
Keywords: Montelukast; Upper respiratory tract infection; leukotriene; Children
MeSH Terms: conditions — Respiratory Tract Infections | interventions — montelukast

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Muntelukast
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Muntelukast — Tablets or granules; 4 mg once a day for 12 weeks
  Other Names: Singulair
  Arms: A
Drug: Placebo — Look alike tablets or granules 1 per day for 12 weeks
  Arms: B

SUMMARY:
Viral upper respiratory tract infection (URI) is one of the most common diseases among toddlers and pre-school children.Complete and effective prevention measures for URI are currently unavailable.

Montelukast (Singulair ) is a selective leukotriene-receptor antagonist that inhibits the cysteinyl leukotriene 1 receptor. It is well tolerated and safe even in young children. Montelukast is an effective treatment for asthma (and allergic rhinitis from 1 year of age. Infections with viruses causing URI such as Influenza A, Rhinovirus and respiratory syncitial virus increases leukotriens levels in nasal secretions. Therefore, one may postulate that leukotriens inhibitors may reduce symptoms during URI. However the effect of montelukast as a treatment for non-specific cough was not properly studied and there are no studies on the effect of montelukast as prevention for URI.

Hypothesis: Prophylactic treatment with Montelukast will reduce the incidence and severity of upper respiratory infection in children.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 to 5 years old without significant health problem.

Exclusion Criteria:

* A previous history of wheezing (requiring treatment with bronchodilators in the last 3 month or more than one treatment in the last year)
* Hospital admission due to reactive air way disease
* Prophylactic use of montelukast or steroids
* Chronic cardiac or respiratory disease
* Presence of acute respiratory tract infection within the 7 days before consideration for the study
* History of allergic Rhinitis
* Children who are receiving chronic medications of any kind
* Known allergy to montelukast
* Inability to get an informed consent from a legal guardian.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The number and duration of URI episodes | 3 month

SECONDARY OUTCOMES:
Severity of URI episodes,number of days with fever,antibiotic and antipyretic usage, unscheduled visits to physicians office, child's absence from day care or kindergarten, parental absence from work, hospital admissions and adverse reaction of the drug. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Mati Berkovitch, MD, Principal Investigator — Assaf-Harofeh Medical Center; Eran Kozer, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (3):
- Israel (3):
  - Kupat Cholim Clalit, Lod
  - Kupat Cholim Clalit, Ramla
  - Assaf Harofeh, Ẕerifin